CLINICAL TRIAL: NCT07161414
Title: A Phase I, Multicenter, Dose Finding and Dose Confirmation Study to Investigate the Pharmacokinetics, and Safety of Subcutaneous Rilvegostomig in Adult Participants With Advanced Solid Tumors Previously Treated With Standard of Care Therapy (ARTEMIDE-subQ)
Brief Title: A Study to Investigate the Pharmacokinetics and Safety of Subcutaneous Rilvegostomig in Adult Participants With Advanced Solid Tumors Previously Treated With Standard of Care Therapy
Acronym: ARTEMIDE-subQ
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D702EC00001; 2025-521614-26-00 (Other: EU CT Number)
Record Dates: First submitted 2025-09-03; First posted 2025-09-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: Recombinant Human Hyaluronidase; Immunooncology monotherapy; T cell Immunoglobulin and Immunoreceptor Tyrosine-based Inhibitory Motif Domain (TIGIT); Programmed Cell Death Protein 1 (PD-1); Bispecific immunotherapy; Checkpoint inhibitor
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (dose finding): Cohort A - SC Rilvegostomig Dose Level 1 (DL1) and rHu (Experimental): Participants will receive IV rilvegostomig (Dose X) as their first dose of study treatment, followed by subsequent treatments with recombinant human hyaluronidase (rHu) and SC rilvegostomig (DL1) at predefined intervals.
  Interventions: Drug: IV Rilvegostomig; Drug: Recombinant Human Hyaluronidase (rHu); Drug: SC Rilvegostomig
- Part 1 (dose finding): Cohort B - SC Rilvegostomig DL2 and rHu (Experimental): Participants will receive IV rilvegostomig (Dose X) as their first dose of study treatment, followed by subsequent treatments with rHu and SC rilvegostomig (DL2) at predefined intervals.
  Interventions: Drug: IV Rilvegostomig; Drug: Recombinant Human Hyaluronidase (rHu); Drug: SC Rilvegostomig
- Part 2 (dose confirmation): SC Rilvegostomig and rHu (Experimental): Participants will receive SC rilvegostomig and rHu.
  Interventions: Drug: SC rilvegostomig + rHu

INTERVENTIONS:
Drug: IV Rilvegostomig — Rilvegostomig administered IV.
  Other Names: AZD2936
  Arms: Part 1 (dose finding): Cohort A - SC Rilvegostomig Dose Level 1 (DL1) and rHu; Part 1 (dose finding): Cohort B - SC Rilvegostomig DL2 and rHu
Drug: Recombinant Human Hyaluronidase (rHu) — rHu administered subcutaneously.
  Arms: Part 1 (dose finding): Cohort A - SC Rilvegostomig Dose Level 1 (DL1) and rHu; Part 1 (dose finding): Cohort B - SC Rilvegostomig DL2 and rHu
Drug: SC Rilvegostomig — Rilvegostomig administered subcutaneously.
  Other Names: AZD2936
  Arms: Part 1 (dose finding): Cohort A - SC Rilvegostomig Dose Level 1 (DL1) and rHu; Part 1 (dose finding): Cohort B - SC Rilvegostomig DL2 and rHu
Drug: SC rilvegostomig + rHu — SC rilvegostomig + rHu administered subcutaneously.
  Arms: Part 2 (dose confirmation): SC Rilvegostomig and rHu

SUMMARY:
The purpose of this study is to determine the subcutaneous (SC) dose that gives rilvegostomig exposure comparable to the intravenous (IV) exposure, and to evaluate the pharmacokinetics (PK) and safety of SC rilvegostomig in adult participants with advanced solid tumors previously treated with standard of care therapy for whom immunooncology (IO) monotherapy would be deemed appropriate by the investigator.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multicenter, multi-part, dose finding and dose confirmation study to evaluate the PK and safety of SC rilvegostomig.

The study includes 2 parts: Part 1 (Dose Finding) and Part 2 (Dose Confirmation).

Part 1 will determine a SC rilvegostomig dose co-administered with rHu that yields drug exposure comparable with IV rilvegostomig. It will include 2 planned dose levels (DL1 in Cohort A and DL2 in Cohort B). Additional dose levels will be added, if needed.

Part 2 will be initiated once a dose has been identified based on Part 1. This part will evaluate the bioavailability, safety, and tolerability of SC rilvegostomig + rHu.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented advanced (metastatic and/or unresectable) solid tumor.
* Participants must have received prior anticancer treatment for the disease under study.
* IO monotherapy deemed appropriate by the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment with no deterioration.
* Minimum life expectancy of ≥ 12 weeks at enrollment.
* Adequate organ and marrow function.
* Body weight ≥ 30 kg.

Exclusion Criteria:

* Any severe or uncontrolled systemic diseases, which makes it undesirable for the participant to participate in the study or that would jeopardize compliance with the protocol.
* History of organ transplant.
* History of another primary malignancy that was active within past 2 years.
* Persistent toxicities caused by previous anticancer treatment(s) excluding alopecia, not yet improved to Grade ≤ 1 or baseline.
* Unstable, symptomatic brain metastasis or spinal cord compression.
* History of leptomeningeal carcinomatosis.
* Active primary immunodeficiency/active infectious disease including tuberculosis (TB), human immunodeficiency virus (HIV) infection or hepatitis A, B or C infection.
* History of clinically significant arrhythmia, cardiomyopathy of any etiology; symptomatic congestive heart failure, history of myocardial infarction within the past 6 months.
* Uncontrolled intercurrent illness including but not limited to ongoing or active known infection; interstitial lung disease (ILD), serious chronic gastrointestinal conditions associated with diarrhea; active non-infectious skin disease requiring systemic treatment.
* Active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.
* Known allergy or hypersensitivity to rilvegostomig, hyaluronidase, or any excipients of the investigational products.
* Participants experienced a toxicity to prior immunotherapy that led to permanent discontinuation of prior immunotherapy.
* Prior anticancer treatment, including immunotherapy, up to 28 days prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-07-19 (Estimated); Study Completion 2029-07-24 (Estimated)

PRIMARY OUTCOMES:
Area under the Concentration-time Curve During One Dosing Interval (AUCtau) | From Day 1 up to end of Cycle 2 in Part 1 and end of Cycle 1 in Part 2 (each cycle will be of 3 weeks)
  Bioavailability based on AUCtau at first SC dose will be determined.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | From Day 1 up to 90 days post last dose (Up to approximately 29 months)
  To assess safety and tolerability of SC rilvegostomig. Safety and tolerability will be evaluated in terms of AEs (graded by CTCAE version 5.0), clinical laboratory assessments, vital signs, physical examinations, and ECOG performance status.
Observed Lowest Concentration before the Next Dose is Administered (Ctrough) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of rilvegostomig (approximately 29 months).
  To assess drug exposure (Ctrough) of SC rilvegostomig comparable to that of IV rilvegostomig.
Average drug concentration over a dosing interval (Cavg) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of rilvegostomig (approximately 29 months).
  To assess drug exposure (Cavg) of SC rilvegostomig comparable to that of IV rilvegostomig.
AUCtau | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of rilvegostomig (approximately 29 months).
  To assess drug exposure of SC rilvegostomig comparable to that of IV rilvegostomig.
Serum rilvegostomig concentration | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of rilvegostomig (approximately 29 months).
  To assess drug exposure (serum concentration) of SC rilvegostomig comparable to that of IV rilvegostomig.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - Research Site, Huntersville, North Carolina
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- United Kingdom (2):
  - Research Site, Newcastle upon Tyne
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/